CLINICAL TRIAL: NCT04920383
Title: An Open-label Study of ALPN-202 Combined With PD-1 Inhibition in Subjects With Advanced Malignancies (NEON-2)
Brief Title: ALPN-202 With PD-1 Inhibition in Advanced Malignancies
Acronym: NEON-2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Alpine Immune Sciences, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIS-B02; MK-3475-D05/KEYNOTE-D05 (Other: Merk Sharp & Dohme LLC)
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Advanced Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): ALPN-202 + pembrolizumab KEYTRUDA®
  Interventions: Drug: ALPN-202; Drug: pembrolizumab KEYTRUDA®

INTERVENTIONS:
Drug: ALPN-202 — Various doses
Drug: pembrolizumab KEYTRUDA® — Varies

SUMMARY:
This is a cohort-based, open-label dose escalation and expansion study in adults with advanced solid tumors or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 to 80 years old at screening
* Pathologically confirmed, locally advanced or metastatic unresectable solid tumor, or Hodgkin or Non-Hodgkin lymphoma (including transformed lymphoma) of an acceptable histology:

  1. that is eligible for treatment with a PD-1 or PD-L1 inhibitor, or
  2. that is refractory or resistant to standard therapy, or
  3. for which standard or curative therapy is not available.
* Have received ≥ 2 prior systemic anti-cancer therapies (lymphoma subjects only)
* Protocol-defined measurable disease
* Available tumor biopsy representative of current disease
* ECOG performance status grade 0-1
* Life expectancy of ≥ 3 months
* Recovery to Grade ≤ 1 for any non-laboratory toxicity resulting from previous anticancer therapy prior to first dose of ALPN-202 (except alopecia, hearing loss, Grade ≤ 2 neuropathy, or endocrinopathy managed with replacement therapy)
* Adequate baseline hematologic, renal, hepatic and cardiac function

Exclusion Criteria:

* Any history of ≥ Grade 3 immune-related adverse event (irAE) requiring discontinuation from treatment or any history of a cardiovascular irAE
* Active or prior pneumonitis or interstitial lung disease
* Presence of any active central nervous system metastases
* Prior organ allograft or allogeneic hematopoietic stem cell transplantation
* Any other serious or uncontrolled health condition, which, in the opinion of the Investigator, would place the subject at undue risk from the study, impair the ability of the subject to receive protocol specified therapy, or interfere with the interpretation of study results.
* Receipt of any protocol-restricted therapy within the timeframes indicated:

  1. Checkpoint inhibitors, including PD-(L)1 (e.g., pembrolizumab, nivolumab, cemiplimab, avelumab, durvalumab), CTLA-4 (e.g., ipilimumab, tremelimumab), and Lag-3 (e.g., relatlimab), costimulatory agonists (including but not limited to CD28, CD134 (OX40), CD137 (4-1BB)): 3 months (135 days for atezolizumab)
  2. Chemotherapy, small molecule anticancer agents (e.g., kinase inhibitors), or radiation: 2 weeks
  3. Other monoclonal antibodies, antibody-drug conjugates, bispecific antibodies, antibody-like drugs, cytokines, cell therapies, or radioimmunoconjugates: 4 weeks
* Any active, known, or suspected autoimmune disease
* Systemic treatment with corticosteroids (> 10 mg/day prednisone) or other immunosuppressive medication
* Any second malignancy active within the previous 3 years
* Active infection requiring therapy at the time of the first dose of ALPN-202.
* Known seropositivity for or active infection by human immunodeficiency virus, hepatitis B or C, or or Severe Acute Respiratory Syndrome Coronavirus 2.
* Known allergies, hypersensitivity, or intolerance to ALPN-202 or excipients in the drug product formulation.
* History of Grade 4 infusion-related, anaphylactic or allergic reaction to any previous Fc-based protein therapy.
* Any serious or uncontrolled cardiovascular condition, including but not limited to:

  1. Any history of myocarditis of any etiology
  2. History of New York Heart Association Class III or IV congestive heart failure, myocardial infarction, unstable angina, cerebrovascular accident, cardiac hospitalization, or other acute uncontrolled heart disease within 6 months of scheduled C1D1
  3. Left ventricular ejection fraction < 45% on screening echocardiogram
  4. Any clinically significant findings on screening EKG such as atrial or ventricular arrythmia (other than sinus tachycardia) or AV conduction abnormality such as left bundle branch block (such subjects may be enrolled after cardiology clearance and Medical Monitor approval)
* Has received prior radiotherapy within 2 weeks of start of study treatment, or have had a history of radiation pneumonitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Dose-limiting Toxicities (DLTs) | Up to 6 weeks following study day 1
  Incidence of DLTs
Adverse Events (AEs) | 30 days after last dose of study drug
  Type, incidence, severity, and seriousness of AEs
Laboratory Abnormalities | Up to 30 days after last dose of study drug
  Type, incidence, and severity of laboratory abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Allison Naumovski, Ph.D., Study Director — Alpine Immune Sciences
Locations (5):
- United States (5):
  - Investigational Site (213), Atlanta, Georgia
  - Investigational Site (212), Boston, Massachusetts
  - Investigational Site (301), Grand Rapids, Michigan
  - Investigational Site (203), Nashville, Tennessee
  - Investigational Site (215), San Antonio, Texas

REFERENCES:
- [Derived] Cavalcante L, Chandana S, Lakhani N, Enstrom A, LeBlanc H, Schmalz J, Lengyel K, Schneider F, Thomas H, Chisamore MJ, Peng SL, Naumovski A, Davar D. Case report of fatal immune-mediated myocarditis following treatment with davoceticept (ALPN-202), a PD-L1-dependent CD28 costimulator and dual PD-L1/CTLA-4 checkpoint inhibitor, in combination with pembrolizumab. J Immunother Cancer. 2024 Aug 13;12(8):e009475. doi: 10.1136/jitc-2024-009475. PMID 39142718
- [Derived] Davar D, Cavalcante L, Lakhani N, Moser J, Millward M, McKean M, Voskoboynik M, Sanborn RE, Grewal JS, Narayan A, Patnaik A, Gainor JF, Sznol M, Enstrom A, Blanchfield L, LeBlanc H, Thomas H, Chisamore MJ, Peng SL, Naumovski A. Phase I studies of davoceticept (ALPN-202), a PD-L1-dependent CD28 co-stimulator and dual PD-L1/CTLA-4 inhibitor, as monotherapy and in combination with pembrolizumab in advanced solid tumors (NEON-1 and NEON-2). J Immunother Cancer. 2024 Aug 3;12(8):e009474. doi: 10.1136/jitc-2024-009474. PMID 39097413